CLINICAL TRIAL: NCT06670365
Title: Evaluating the Efficacy of Heat Acclimation by Warm Water Immersion for Mitigating Hyperthermia and Cardiovascular Demand in Older Adults During Indoor Overheating.
Brief Title: Enhancing Heat Resiliency in Older Adults During Indoor Overheating Via Heat Acclimation by Warm Water Immersion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Glen P. Kenny, Professor, University of Ottawa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HEPRU-2024-09-A
Record Dates: First submitted 2024-10-29; First posted 2024-11-01 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Hyperthermia; Thermoregulation; Aging; Heat Acclimation and Thermotolerance
Keywords: thermoregulation; heat illness; heat acclimation; extreme heat events; women; indoor overheating; water immersion
MeSH Terms: conditions — Hyperthermia; Heat Stress Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daylong exposure to indoor overheating (Experimental): Prior to and following the warm-water immersion protocol, participants will undergo a 10-hour passive heat exposure where they will remain in a climate-controlled chamber regulated at 36°C and 45% humidity (temperatures experienced indoors during extreme heat events in North America). During this time they will remain seated with the exception of hourly 5-minute breaks to stretch.
  Interventions: Other: Heat acclimation by warm-water immersion

INTERVENTIONS:
Other: Heat acclimation by warm-water immersion — Participants will be immersed in a whirlpool tub to the shoulder level in a circulated water bath maintained at ~40°C until their core temperature achieves a steady-state of 38.5°C for 60 minutes. The warm-water immersion protocol will be repeated for 6 more consecutive days.

SUMMARY:
As overheating in buildings is expected to increase as global warming continues, proactive measures to increase heat resiliency in heat-vulnerable older people are needed, especially for those without access to home cooling or reliable sources of electricity. While short-term heat acclimation through exercise in the heat has been shown to increase heat dissipation and decrease both the physical and mental stress imposed on individuals exposed to heat, such protocols are not tenable for older, sedentary adults. A recent report showed that seven consecutive days of warm-water immersion improved whole-body heat loss and reduced physiological strain as assessed during an exercise-heat stress in habitually active older men This represents a critical finding as an increase heat-loss capacity would serve as an important safeguard for older adults exposed to indoor overheating due to lack of air-conditioning. While this preliminary data highlights passive hot water immersion as a promising strategy for increasing heat-resilience in vulnerable adults, work is needed to confirm its efficacy in more "real-world" environments. Thus, this study aims to assess the effectiveness of a 7-day passive heating (warm-water immersion with core temperature clamped at ~38.5°C for the final 60 minutes) protocol in mitigating increases in thermal and cardiovascular strain in older females exposed to daylong (10-hours) indoor overheating (36°C, 45% relative humidity) prior to and following the passive heating intervention. Relative to males, females have a reduced heat loss capacity (~5%), which is driven by differences in the activation of heat loss responses (i.e., skin blood flow and sweating). Although there have been mixed findings with regards to the influence of sex as a mediating factor for heat-related mortality, some studies suggest that females are at a higher risk of heat-related mortality and morbidity compared to males, especially amongst older individuals (≥65 years). Notably, a greater proportion of older females died compared to their male counterparts during the 2021 Western Heat Dome. While the underlying causes for these differences remain unclear, greater cardiovascular strain may place females at higher mortality risk during extreme heat.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking.
* English or French speaking.
* Ability to provide informed consent.
* With or without a) chronic hypertension (elevated resting blood pressure; as defined by Heart and Stroke Canada and Hypertension Canada), b) type 2 diabetes as defined by Diabetes Canada, with at least 5 years having elapsed since time of diagnosis

Exclusion Criteria:

* Episode(s) of severe hypoglycemia (requiring the assistance of another person) within the previous year, or inability to sense hypoglycemia (hypoglycemia unawareness).
* Serious complications related to your diabetes (gastroparesis, renal disease, uncontrolled hypertension, severe autonomic neuropathy).
* Uncontrolled hypertension - BP >150 mmHg systolic or >95 mmHg diastolic in a sitting position.
* Restrictions in physical activity due to disease (e.g. intermittent claudication, renal impairment, active proliferative retinopathy, unstable cardiac or pulmonary disease, disabling stroke, severe arthritis, etc.).
* Use of or changes in medication judged by the patient or investigators to make participation in this study inadvisable.
* Cardiac abnormalities identified during screening

Ages: 65 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Core temperature (Peak) during daylong heat exposure | End of 10 hour daylong heat exposure
  Peak rectal temperature (15 min average) during exposure. Rectal temperature is measured continuously throughout the 10 hours of the simulated heat wave performed prior to and following the 7-day heat acclimation by warm-water immersion.
Core temperature (AUC) during daylong heat exposure | End of 10 hour daylong heat exposure
  Area under the curve (AUC) of rectal temperature (in degree-hours) during the 10 hour simulated heat wave exposure performed prior to and following the 7-day heat acclimation by warm-water immersion.
Heat rate (Peak) during daylong heat exposure | End of 10 hour daylong heat exposure
  Peak Heart rate (15-min average) during the 10 hour simulated heat wave exposure performed prior to and following the 7-day heat acclimation by warm-water immersion.
Heat rate (AUC) during daylong heat exposure | End of 10 hour daylong heat exposure
  Area under the curve (AUC) of heart rate during the 10 hour simulated heat wave exposure performed prior to and following the 7-day heat acclimation by warm-water immersion.
Cardiac response to standing from supine (30:15 Ratio) during daylong heat exposure | At the start (hour 0) and end of daylong heat exposure (hour 10)
  Cardiac response to standing evaluated as the ratio between the highest R-wave to R-wave interval (lowest heart rate) measured at the 30th heart beat after standing from supine (+/- 5 beats) and the lowest R-wave to R-wave interval (highest heart rate) measured at the 15th heart beat after standing (+/- 5 beats). Cardiac response to standing will be evaluated twice, during two lying-to-standing tests (separated by 10 min of supine rest).
Systolic Response to Standing From Supine during daylong heat exposure | At the start (hour 0) and end of the daylong heat exposure (hour 10)
  Systolic blood pressure response to standing evaluated as the difference in blood pressure measured between the standing and supine. Standing systolic blood pressure will be taken as the lowest value of those measured after 60 and 120 seconds of standing. Systolic response to standing will be evaluated twice, during two lying-to-standing tests (separated by 10 min of supine rest). Assessed at the start and end of the 10 hour simulated heat wave exposure performed prior to and following the 7-day heat acclimation by warm-water immersion.
Heart rate variability: RMSSD during daylong heat exposure | At the start (hour 0) and end of the daylong heat exposure (hour 10)
  Root mean squared standard deviation of normal-to-normal R-wave to R-wave intervals (RMSSD) measured during 5 minutes of paced breathing (15 breaths/min) with participants in the supine position. RMSSD will be evaluated twice, during two paced breathing periods (separated by 4 min of supine rest).
Heart rate variability: SDNN during daylong heat exposure | At the start (hour 0) and end of daylong heat exposure (hour 10)
  Standard deviation of normal-to-normal R-wave to R-wave intervals (SDNN) measured during 5 minutes of paced breathing (15 breaths/min) with participants in the supine position. SDNN will be evaluated twice, during two paced breathing periods (separated by 4 min of supine rest).
Thermal comfort scale during daylong heat exposure | End of 10 hour daylong heat exposure
  Thermal comfort assessed via a visual analog scale ranging from extremely uncomfortable to extremely comfortable (midpoint: neutral).
Thirst sensation scale during daylong heat exposure | End of 10 hour daylong heat exposure
  Thirst sensation scale assessed via a visual analog scale (9: very, very thirsty to 1: Not thirsty at all)
Thermal sensation scale during daylong heat exposure | End of 10 hour daylong heat exposure
  Thermal sensation assessed via a visual analog scale ranging from extremely hot to neutral (midpoint: hot).
Arousal scale during daylong heat exposure | End of 10 hour daylong heat exposure
  Felt arousal scale assessed via a visual analog scale ("How worked up are you?") ranging from "high arousal" to "low arousal".
Fluid loss during daylong heat exposure | End of 10 hour daylong heat exposure
  Body fluid loss calculated as a change in body weight from pre-exposure values (corrected for food intake and deification).
Fluid consumption during daylong heat exposure | End of 10 hour daylong heat exposure
  Average hourly fluid consumption calculated by weighing participant water intake at the start and end of each hour of exposure (normalized to the exposure duration).
Changes in plasma volume during daylong heat exposure | End of 10 hour daylong heat exposure
  Change in plasma volume from baseline values calculated from duplicate measurements of hemoglobin and hematocrit at the start and end of each exposure using the technique by Dill and Costill
Systolic blood pressure during daylong heat exposure | End of 10 hour daylong heat exposure
  Systolic blood pressure measured in triplicate via automated oscillometry (~60 seconds between measures)
Diastolic blood pressure during daylong heat exposure | End of 10 hour daylong heat exposure
  Diastolic blood pressure measured in triplicate via automated oscillometry (~60 seconds between measures)
Systolic Response to Standing From Supine during daylong heat exposure | End of 10 hour daylong heat exposure
  Systolic blood pressure response to standing evaluated as the difference in blood pressure measured between the standing and supine. Standing systolic blood pressure will be taken as the lowest value of those measured after 60 and 120 seconds of standing. Systolic response to standing will be evaluated twice, during two lying-to-standing tests (separated by 10 min of supine rest).
Rate pressure product during daylong heat exposure | At the start (hour 0) and end of the daylong heat exposure (hour 10)
  Rate pressure product, an index of myocardial work and strain, calculated as systolic blood pressure x heart rate.
Orthostatic intolerance symptoms assessment during daylong heat exposure | End of 10 hour daylong heat exposure
  Cumulative sum of scores on 6 questions asking participant to rank symptoms associated with orthostatic intolerance during the lying to standing tests. All symptoms scored on a scale from 0 (none) to 10 (worst possible) and include feelings of: (1) "dizziness, lightheadedness, feeling faint, or feeling like you might black out"; (2) "Problems with vision (blurring, seeing spots, tunnel vision, etc.)"; (3) "Weakness"; (4) "Fatigue"; (5) "Trouble concentrating"; and (6) "Head and neck discomfort".
Reaction time (cognitive function) during daylong heat exposure | At the start (hour 0) and end of the daylong heat exposure (hour 10)
  Participants will be provided with a tablet device with the Sway Medical testing platform for the assessment of reaction time. Participants will be asked to initiate a movement of the device in response to a visual cue.
Impulse control (cognitive function) during daylong heat exposure | At the start (hour 0) and end of the daylong heat exposure (hour 10)
  Participants will be provided with a tablet device with the Sway Medical testing platform for the assessment of impulse control. Participants will be asked to respond to both "go" and "no-go" visual cues. In response to the "go" cue, participants will initiate a movement of the device.
Memory recall (cognitive function) during daylong heat exposure | At the start (hour 0) and end of the daylong heat exposure (hour 10)
  Participants will be provided with a tablet device with the Sway Medical testing platform for the assessment of memory recall. Participants complete both a delayed recall test and a working memory test.
CDC 4-Stage Balance Test (Postural stability) during daylong heat exposure | At the start (hour 0) and end of the daylong heat exposure (hour 10)
  To assess postural stability, participants hold a tablet to their chest, then auditory cues guide participants through four consecutive stances, feet side by side, instep of one foot touching the big toe of the other foot, tandem stand with one foot in front of the other, heel touching toe, and stand on one foot. The balance assessment will be evaluated based on movement detected by an accelerometer integrated into the hardware of the tablet device (Sway Medical Inc).
BTrackS Balance Assessment (Postural stability) during daylong heat exposure | At the start (hour 0) and end of the daylong heat exposure (hour 10)
  To assess postural stability, participants will be asked to stand on a BTracks force plate with their feet spread out to shoulder width, hand on their hips and eyes closed. The assessment will comprise of four trials (one practice trial) lasting 20 seconds in length and 20 seconds between trials. Center of pressure (COP) vector data along vertical (y) and horizontal (x) axes will be summed for the total path excursion length (cm) during each trial.

SECONDARY OUTCOMES:
Muscle oxygen during battery of cardiovascular, cognition and postural stability tests during daylong heat exposure | At the start (hour 0) and end of the daylong heat exposure (hour 10)
  Participants will be attached with 2 probes to measure tissue oxygenation on two locations via a non-invasive tool: near-infrared spectroscopy (NIRS). The device (Portalite, Artinis Medical, The Netherlands) is placed on the left prefrontal cortex and muscle belly of the vastus lateralis. The change in tissue oxygenation at both sites will be assessed as a percent change from baseline.
Profiles of Mood States (POMS) during daylong heat exposure | At the start (hour 0) and end of the daylong heat exposure (hour 10)
  Potential changes in mood (7 subscales of mood: tension, anger, depression, fatigue, confusion, vigor and esteem-related affect). The POMS-40 is a validated, self-administered questionnaire that examines seven distinct aspects of mood state across two positive subscales (Esteem-Related Affect, and Vigor) and five negative subscales (Fatigue, Tension, Confusion, Anger, and Depression), which are described across 40 distinct adjectives (reference). For each individual item, participants were asked to describe "how you feel right now" by responding using a 5-point Likert scale (0 = "Not at all", 1 = "A little", 2 = "Moderately", 3 = "Quite a lot", or 4 = "Extremely"). The values of items associated with a specific subscale (e.g., Fatigue) were summed to calculate its score.
Environmental Symptoms Questionnaire (ESQ) | At the start (hour 0) and end of the daylong heat exposure (hour 10)
  Self-reported environmental reactions and medical symptomatology associated with prolonged heat exposure. The ESQ-IV is a validated 68-item, self-administered questionnaire that has been used successfully in identifying symptomatology during exposure to a wide variety of environmental conditions, including heat exposure [24, 25]. Participants are asked to assess and described "how you have been feeling today" by responding to each item using a 6-point Likert scale (0 = "Not at all", 1 = "Slight", 2 = "Somewhat", 3 = "Moderate", 4 = "Quite a bit", or 5 = "Extreme"). Total Symptom Score was calculated from this data by taking the sum of the intensity ratings from all 68 individual items using reverse scores for the three positive items from the list ("I Felt Good", "I Felt Alert", and "I Felt Wide Awake").
Sleepiness during daylong heat exposure A | End of 10 hour daylong heat exposure
  Karolinska sleepiness scale measures the subjective level of sleepiness at a particular time during the day on a scale of 1 to 10. 1 = extremely alert and 10 = extremely sleepy
Sleepiness during daylong heat exposure B | End of 10 hour daylong heat exposure
  Stanford sleepiness scale consists of only one item, where participant must identify one of seven statements that best represents their level of perceived sleepiness. It employs a scale of 1 to 7 with 1 = feeling wide awake and 7 = sleep onset soon

CONTACTS AND LOCATIONS:
Overall Officials: Glen P Kenny, PhD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be made available with approved analysis plan and signed access agreement
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Following publication of the main study report(s)
Access Criteria: Approved analysis plan and signed access agreement